CLINICAL TRIAL: NCT00338468
Title: An Open-Label Pilot Study to Assess Disability in Anemic Elderly Patients With Chronic Kidney Disease Receiving PROCRIT (Epoetin Alfa)
Brief Title: A Study to Assess Disability in Anemic Elderly Patients With Kidney Disease Receiving PROCRIT (Epoetin Alfa)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was stopped early due to slow enrollment.
Sponsor: Ortho Biotech Products, L.P. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004606
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-03

CONDITIONS: Anemia; Kidney Diseases
Keywords: Anemia; Elderly; Hemoglobin level; Chronic Kidney Disease
MeSH Terms: conditions — Anemia; Kidney Diseases; Renal Insufficiency, Chronic | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to assess disability in anemic patients over the age of 65 who have kidney disease and are receiving weekly PROCRITÂ® (Epoetin Alfa, a glycoprotein that stimulates red blood cell production).

DETAILED DESCRIPTION:
This is an open-label study in which PROCRIT® (Epoetin Alfa) will be given on a weekly basis starting at a dose lower than is currently approved by the U.S. FDA because treatment is beginning at a higher hemoglobin than usual. There is recent evidence to suggest that problems with disability occur in persons over 65 at higher hemoglobins than previously recognized. Currently, PROCRIT® (Epoetin Alfa) is prescribed for patients with chronic kidney disease three times a week at a dose of approximately 5,000 and 10,000 units per injection depending on the patient's weight. This study is starting with a lower dose because treatment is beginning earlier than it normally would. Currently, doctors usually do not begin PROCRIT® (Epoetin Alfa) in patients with chronic kidney disease until their hemoglobin is <10 g/dL.

In this study PROCRIT® (Epoetin Alfa) will be given on a weekly basis starting at 5,000 units per injection if hemoglobin is <12 g/dL. Each week hemoglobin will be checked and if after four weeks of treatment it is < 13 g/dL, the PROCRIT® (Epoetin Alfa) dose will be increased to 10,000 Units. After another four weeks of treatment if the hemoglobin is <13 g/dL, PROCRIT® (Epoetin Alfa) will be increased to 20,000 units. After another four weeks of treatment if the hemoglobin is <13 g/dL, PROCRIT® (Epoetin Alfa) will be increased once more to a final dose of 40,000 units. In this study, patients will be treated with doses higher than currently approved for patients with chronic kidney disease. The primary measures of efficacy will be assessed using two disability tests to measure physical function compared from baseline to Week 5, Week 9, Week 13, Week 17/ Early Withdrawal and Week 20/Follow-up. The first test is called the "Short Physical Performance Battery" (SPP) which will test how well someone sits, stands and walks. The second test is called the "Six Minute Walk Test" (6MWT) which measures how far someone can walk during a six-minute period. Normal walking aids are allowed during this test. The study will also evaluate hemoglobin levels, number of transfusions, safety, incidence of anti-erythropoietin antibodies, Quality of Life and cognitive function (a measure of how clearly one is thinking). The study hypothesis is that physical function will improve when the hemoglobin level is increased. Patients will receive PROCRIT® (Epoetin Alfa) on a weekly basis starting at 5,000 units per injection (up to a maximum of 40,000 units).

ELIGIBILITY:
Inclusion Criteria:

* Patients having chronic anemia and chronic renal failure
* have lessened physical function
* be community dwelling (defined as not admitted to an assisted nursing facility, nursing home or hospital at the time of enrollment. An assisted nursing facility is considered any living situation where daily care is being provided by recognized health care professionals from that facility.)

Exclusion Criteria:

* History of bacterial infection requiring hospitalization and intravenous antibiotics or transfusion within 1 month prior to enrollment
* anemia due to iron, folate, or vitamin B12 deficiency
* gastrointestinal bleeding
* anticipated to begin dialysis within 4 months following enrollment into the study
* History of thrombotic disease within the past 3 months, or on anticoagulation therapy at enrollment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-11; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Change in physical function score as measured by the Six Minute Walk Test (6MWT) and Short Physical Performance (SPP) Summary Score compared from Baseline to Week 5, Week 9, Week 13, Week 17/ Early Withdrawal and Week 20/Follow-up.

SECONDARY OUTCOMES:
Proportion of patients who achieve the target hemoglobin levels of > 13.0 g/dL and < =14.0 g/dL (independent of transfusion within 1 month of assessment) compared from Baseline to Week 5, Week 9, Week 13, Week 17/ Early Withdrawal and Week 20/Follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ortho Biotech Products, L.P. Clinical Trial, Study Director — Ortho Biotech Products, L.P.

REFERENCES:
- See also: An Open-Label Pilot Study to Assess Disability in Anemic Elderly Patients with Chronic Kidney Disease Receiving PROCRIT (Epoetin alfa) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=924&filename=CR004606_CSR.pdf